CLINICAL TRIAL: NCT06634030
Title: A Randomized, Double-Blinded, Controlled Trial Evaluating Recombinant Human Platelet-Derived Growth Factor B (rhPDGF-BB)-Enhanced Wound Matrix in the Reconstruction of Full-Thickness Head or Neck Defects Following Skin Cancer Excision
Brief Title: Evaluating rhPDGF-BB-Enhanced Wound Matrix for Head and Neck Reconstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Lynch Regenerative Medicine, LLC (Unknown)
Responsible Party: Principal Investigator, Wesley Thayer, Vice Chair of Research, Department of Plastic Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 240597
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Wound Healing; Surgical Wound; Graft Failure
Keywords: Complex Surgical Defect; Skin Cancer Excision; Platelet-Derived Growth Factor; Skin Graft
MeSH Terms: conditions — Surgical Wound | interventions — Becaplermin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline matrix (Placebo Comparator): Participants receive wound matrix saturated with normal saline.
  Interventions: Drug: Saline
- rhPDGF-BB matrix (Experimental): Participants receive wound matrix saturated with rhPDGF-BB.
  Interventions: Drug: RhPDGF-BB

INTERVENTIONS:
Drug: RhPDGF-BB — 0.3 mg/mL rhPDGF-BB
  Arms: rhPDGF-BB matrix
Drug: Saline — Normal saline
  Arms: Saline matrix

SUMMARY:
Skin cancers such as basal cell carcinoma (BCC), squamous cell carcinoma (SCC), and melanoma lesions that develop on the head and neck are treated by Mohs surgery or wide local excision to remove all tumor cells and preserve the normal tissue. These surgical techniques may result in large wounds requiring reconstructive surgery to restore function and aesthetics. Older, frail patients are particularly vulnerable to complications from these invasive procedures often leaving them to care for chronic wounds until a split-thickness skin graft can be placed. Recombinant human platelet-derived growth factor (rhPDGF) is a manufactured protein that signals through the PDGF receptor, PDGFRβ, to mediate inflammation, granulation, angiogenesis, and remodeling during wound healing and skin repair and is FDA-cleared for diabetic neuropathic ulcers and periodontal bone and soft tissue reconstructions. Preclinical and clinical data suggest that rhPDGF may be a viable therapeutic strategy to augment the reconstruction of these complex surgical wounds by accelerating healing and reducing the time-to-readiness for skin graft placement.

DETAILED DESCRIPTION:
This Phase II clinical trial will evaluate the potential efficacy of rhPDGF-BB-enhanced wound matrix versus wound matrix saturated with normal saline to augment the reconstruction of head and neck defects that cannot approximate and heal by primary intention following skin cancer excision. This prospective, double-blinded, single-site study will randomize participants into two arms - intervention and control - comparing the granulation rates of the wound bed, skin graft success, aesthetic outcomes, and quality of life. After recruiting, consenting, and screening, participants will be scheduled for the baseline procedure to place the wound matrix into the wound bed. Randomization will occur the day of the procedure, and both the investigator and participant will be blinded. To achieve balance in treatment allocation, randomization blocks of 4 (2 interventions : 2 controls) will be stratified by anatomical location, scalp versus face/neck, and greatest dimension, < or = 3cm versus > 3cm, of the surgical defect.

Following the baseline procedure, participants will return for their first follow-up visit on day six for a clinical examination, suture removal, and wound dressing change, and follow-up visits will occur weekly for 8 weeks thereafter. At each visit, participants will complete the VAS pain scale and discuss any adverse events, the wound will be photographed and examined, and the investigator will assess the percent granulation and readiness for a skin graft. Participants will also submit daily photos of the wound while performing dressing changes at home starting on day seven until the skin graft procedure is completed. These photographs will be taken using a wound imaging application capable of ensuring a quality image, measuring the area of the wound, and transfer of the images to password-protected, cloud-based storage. The images will be analyzed by blinded wound experts, retrospectively, to determine the precise day (rather than the week) that the wound bed achieved 95-100% granulation. Placement of the skin graft may occur anytime between the first follow-up visit 1 week after the baseline procedure through 8 weeks. After the skin graft is placed, participants will continue the weekly visits through 8 weeks following the baseline procedure to assess pain and graft take. Under routine care with a wound matrix (no rhPDGF-BB), the average time to readiness is 4-6 weeks in this patient population. Here, we aim to reduce the time to readiness by adding rhPDGF-BB.

ELIGIBILITY:
Inclusion Criteria:

* Underwent surgery to completely remove skin cancer, either Mohs micrographic or wide local excision, that left a full-thickness surgical defect of the head or neck measuring between 1.5-10cm in greatest dimension with clear margins as assessed in the pathology report.
* Margins of the wound cannot be approximated or closed with stitches, sutures, staples, or glue
* Surgeon does not plan for immediate skin graft or flap
* Aged >21 years old
* Willing and able to provide informed consent for study participation and compliance with study protocol
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Medical conditions that would, in the opinion of the Investigator or treating provider, compromise the safety of the individual with study participation and/or the ability of the individual to follow study protocol
* The device will not fit the contour of the base of the wound bed
* Evidence of current clinical infection as demonstrated by the invasion of bacteria into the healthy viable tissue on the periphery of the wound (colonization of wound bed due to normal flora or environment is not exclusionary)
* Prior radiation therapy at the application site
* Known allergic reactions to porcine tissue, porcine collagen, or yeast-derived products
* Currently enrolled in a drug or device trial or within 30 days of last investigational drug or device administration at baseline visit where investigational treatment (drug or device) was placed in wound bed or may potentially interact with study treatment
* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time-to-Readiness for Skin Graft in Days | Daily, starting at day 7 up to day 56 following the baseline procedure
  Time-to-readiness of the wound for a skin graft as determined by clinical review of wound bed granulation in photographic images taken daily starting at day 7 following the baseline procedure.

SECONDARY OUTCOMES:
Granulation Rate | Daily, starting at day 7 up to day 56 following the baseline procedure
  Percent granulation versus time in days as determined by clinical assessment of the percent granulation of the wound bed in photographic images taken daily starting at day 7 following the baseline procedure.
Change in Granulation on a 5-Point Scale | Weekly, starting at week 1 up to week 8 following the baseline procedure
  Weekly ordinal scale outcomes of granulation as determined by clinical assessment of the percent granulation of the wound bed in photographic images taken daily starting at day 7 following the baseline procedure. Ordinal scale ranges from 1 to 5 in the increments below.
  * 0-25% granulation = 1
  * 26-50% granulation = 2
  * 51-75% granulation = 3
  * 76-95% granulation = 4
  * Ready for a skin graft = 5
Time-to-Readiness for Skin Graft in Weeks | Weekly, starting at week 1 up to week 8 following the baseline procedure
  Time-to-readiness of wound for a skin graft as assessed by clinical examination at routine care, post-surgery, weekly visits.
Time to Skin Graft in Days | From day 7 up to day 566 following the baseline procedure
  Time in days to skin graft procedure completed following the baseline procedure
Percentage of Skin Graft Take | Week 1 following skin graft placement
  Skin graft take (percent graft take) as assessed by clinical examination at routine care, post-surgery visit at week 1 after the grafting procedure.
Aesthetics Rating at Week 8 | Week 8
  Aesthetics rating of the wound as assessed by clinical examination at the final week 8 follow-up visit using an ordinal scale from 0 (very ugly) to 10 (very nice).
Scar Scale at Week 8 | Week 8
  Scar rating of the wound as assessed by clinical examination at the final week 8 follow-up visit, with rating determined by the rankings of seven wound qualities on an ordinal scale from 1 (normal skin) to 10 (worst scar imaginable).
Change from Baseline in Pain on an 11-Point Scale | From enrollment through week 8
  Weekly self-reported participant surveys will assess average pain intensity on an 11-point scale. Possible scores range from 0 (No Pain) to 10 (Worst Pain).
Change from Baseline in Quality of Life | From enrollment through week 8
  Change in quality of life based on a self-reported 12-question survey taken at baseline and at week 8.
Number of Participants Recruited and Eligible | Monthly up to month 15
  Total number of participants that were recruited and eligible for the study.
Number of Participants Randomized Per Month | Monthly up to month 15
  Number of participants that were randomized each month of the study.
Proportion of Participants Retained at Week 8 | Week 8
  Proportion of participants retained in the study at week 8 (end of study).
Weekly Percentage of Completed Daily Photos at Week 8 | Weekly, week 1 up to week 8
  Participant adherence to daily wound photograph schedule.
Concordance of Time-to-Readiness Between Photograph Assessments versus Clinical Exams | Weekly, week 1 up to week 8
  Weekly concordance of time-to-readiness assessed by photographs vs. time-to-readiness assessed by clinical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley P Thayer, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided